CLINICAL TRIAL: NCT00593879
Title: A Multi-Center, Double Blind, Randomized, Placebo-Controlled, Parallel Group, Flexible Dose Titration, Add-On Study of Mecamylamine 5.0 to 10 mg, in the Treatment of Major Depressive Disorder With Subjects Who Are Partial or Non- Responders to Citalopram Therapy.
Brief Title: Flexible Dose Titration Add-on Study to Treat Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Geoffrey Dunbar, VP Clinical Development & Regulatory Affairs, Targacept, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-5231-023-CRD-003
Record Dates: First submitted 2007-12-19; First posted 2008-01-15 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Major Depressive Disorder
Keywords: MDD; Depression; Mecamylamine; Add-on Therapy; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Mecamylamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): Placebo
  Interventions: Drug: Mecamylamine
- 2 (Experimental)
  Interventions: Drug: Mecamylamine

INTERVENTIONS:
Drug: Mecamylamine — 2.5mg mecamylamine Hcl, tablet form taken twice a day (total of 5.0mg). For 7.5 mg dose group, 2 tablets taken morning, one tablet evening. At 10.0mg, 2 tablets taken twice daily.
  Other Names: Inversine

SUMMARY:
Depressed patients will receive 6 weeks of citaloprma (20-40mg) therapy. Subjects who have an inadequate response (partial or non-responder) will be randomized to receive either mecamylamine (5-10mg) or placebo added to their citalopram for a further 8 weeks.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo controlled, parallel group, flexible dose titration, add-on study. Male or female subjects aged 18-70 years suffering from Major Depressive Disorder according to DSM-IV, with a HAMD-17 score greater than 21 and a CGI-Severity of Illness score greater or equal to 4, will be started on open labeled citalopram treatment. The dose of citalopram may be increased form 20mg to 40mg over a six week period, depending on investigator assessment of tolerability and efficacy. At the end of this treatment, subjects with a HAMD-17 score greater or equal to 14 and a CGI-Severity of Illness score greater or equal to 4 will be considered as partial or non-responders and will be entered into the double blind phase of the study. Subjects will be randomized to either mecamylamine or placebo for a further 8 weeks. Citalopram medication will remain constant while mecamylamine (or placebo) can be increased from 5.0 to 7.5 to 10.0mg based on investigator assessment of tolerability and efficacy.

Plasma samples for citalopram assay will be collected at the start and end of the double blind phase to exclude any mecamylamine effect being due to a drug:drug interaction.

Approximately 500 subjects will be entered into the open-label phase of the study and approximately 160 into the double blind phase. The study will be conducted in India and the USA.

ELIGIBILITY:
Inclusion Criteria:

(A) Open Phase

* Male or female subjects aged 18-70 years.
* Diagnosis of major depressive disorder (MDD) according to DSM-IV and confirmed via MINI diagnostic scale.
* Able to give written informed consent.
* HAMD-17 score greater than 21.
* CGI-Severity of Illness score greater than or equal to 4.
* No clinically significant abnormality on physical examination, vital signs, ECG or laboratory tests (biochemical, hematological, urinary) at screening.
* Women of child bearing potential with a negative urine pregnancy test and willing to use acceptable methods of contraception.

(B)Double Blind Phase:

* Subjects still to meet DSM-IV criteria for MDD.
* Subjects continue to meet all of the inclusion and exclusion criteria.
* HAMD-17 score greater than or equal to 14.
* CGI severity of illness score greater than or equal to 4.
* Women of child bearing potential with a negative urine pregnancy test and willing to use acceptable methods of contraception.

Exclusion Criteria:

* Aged below 18 years and above 70 years.
* Failure to meet DSM IV criteria for MDD.
* HAMD-17 less than or equal to 21 (open-label phase only).
* CGI Severity of Illness score less than 4.
* Clinically significant changes in physical examination, vital signs, ECG or laboratory tests at screening.
* Any other co morbid psychiatric illness confirmed by MINI diagnostic scale, especially bi-polar disorder, schizophrenia or dementia.
* Subjects with significant suicidal risk upon clinical assessment.
* Subjects who have treatment resistant depression i.e. who have failed adequate course (daily dose and duration of treatment) of one or more antidepressants.
* History of alcohol or drug abuse over the last 6 months.
* History of seizures or seizure disorders.
* Seropositive for HIV or hepatitis B (antibody or antigen).
* Any other severe progressive and uncontrolled medical condition.
* For controlled other medical conditions, medication to be unchanged over the 2 months preceding screening, or else the patient will be excluded.
* Subjects with Glaucoma, Kidney Disease or Heart Disease.
* Known hypersensitivity to mecamylamine.
* Women of child bearing potential not taking adequate contraception and women breastfeeding.
* Other investigational drug in previous 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-02; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
HAMD-17 group mean change from baseline to endpoint and/or the proportion of subjects considered to be full responders or in remission with a HAMD-17 score less than or equal to 7 at the end of treatment. | 8 weeks

SECONDARY OUTCOMES:
Montgomery Asbery depression rating sclae, Clinical Global Impression Scale - Severity, Clinical Global Impression Sacle - Change, Sheehan irritability scale, Sheehan disability scale | 8 weeks
Blood biochemistry, urnie analysis, blood pressure, heart rate, ECG | 8 weeks
Citalopram plasma bloods at week 6 and 14. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Dunbar, MD, Study Director — Targacept Inc.